CLINICAL TRIAL: NCT03301740
Title: Ultrafiltration Profiling and Outcomes Among Individuals on Maintenance Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-1057; 1K23DK109401 (NIH)
Record Dates: First submitted 2017-09-21; First posted 2017-10-04 (Actual); Results first posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2019-01

CONDITIONS: End Stage Renal Disease
Keywords: Ultrafiltration profiling; Hemodialysis; Dialysis; Cardiovascular outcomes; Patient-reported outcomes; Crossover study design; End Stage Renal Disease; Ultrafiltration; Echocardiogram; Blood pressure; Hypotension; Symptoms
MeSH Terms: conditions — Kidney Failure, Chronic; Hypotension

STUDY DESIGN:
Intervention Model Description: The study is a 4-phase crossover trial in which participants are successively alternated between conventional HD and conventional HD + linear UF profiling across 4 phases with intervening wash-out periods. The study compares conventional HD (the participant's standard HD prescription with no UF profiling) to conventional HD + linear UF profiling. Participants will be randomly allocated to conventional HD or conventional HD + linear UF profiling for phase 1. Participants will undergo 9 treatments during each phase for a total of 18 conventional HD treatments and 18 UF profiled treatments. Participants will undergo 3 wash-out HD treatments between phases.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be double-blinded in that participants will not be informed of the treatment paradigm. Investigators, including those performing transthoracic echocardiography (TTE) interpretation, will be blinded to treatment paradigm. Ultrasonographers performing intra-HD TTEs will be blinded to treatment paradigm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UF Profiling Phase First (Experimental): First treatment phase begins with linear UF profiling during HD.
  Participants randomized to starting with the experimental UF profiling phase will receive 9 HD treatments with UF profiling (1st experimental phase). Following a 3 conventional HD treatment wash-out period, participants will then cross over to 9 conventional HD treatments (1st control phase). Following a 2nd 3 conventional HD treatment wash-out period, participants will cross over to 9 HD treatments with UF profiling (2nd experimental phase). Following a 3rd conventional HD treatment wash-out period, participants will cross over to 9 conventional HD treatments (2nd control phase).
  Interventions: Other: UF profiling during HD; Other: Conventional HD
- Conventional HD Phase First (Experimental): First treatment phase begins with conventional HD.
  Participants randomized to starting with the control conventional HD phase will receive 9 conventional HD treatments (1st control phase). Following a 3 conventional HD treatment wash-out period, participants will then cross over to 9 HD treatments with UF profiling (1st experimental phase). Following a 2nd 3 conventional HD treatment wash-out period, participants will cross over to 9 conventional HD treatments (2nd control phase). Following a 3rd conventional HD treatment wash-out period, participants will cross over to 9 HD treatments with UF profiling (2nd experimental phase).
  Interventions: Other: UF profiling during HD; Other: Conventional HD

INTERVENTIONS:
Other: UF profiling during HD — Experimental arm: Linear UF profiling (linearly decreasing UF rate with a UF rate starting at 1.33 times the rate that would be needed at a constant UF rate to achieve the desired post-weight; pre-programmed "profile 2" on a Fresenius 2008K machine, the machine used in all participating clinics). Ultrafiltration profiling will be performed using Fresenius 2008K dialysis machines in accordance with manufacturer instructions.
Other: Conventional HD — Control arm: Conventional HD (routine care) is the participant's standard HD prescription without UF profiling.

SUMMARY:
The rate of fluid removal (ultrafiltration, UF) during hemodialysis (HD) may contribute to cardiovascular morbidity and mortality among individuals receiving maintenance HD. More rapid UF rates are associated with higher morbidity and mortality. Ultrafiltration profiling, the practice of varying UF rates to maximize fluid removal during periods of greatest hydration and plasma oncotic pressures, is one treatment modification that may reduce UF-related harm without necessitating reduction in interdialytic fluid intake or longer HD treatments. To date, UF profiling has not been adequately studied independent of sodium profiling.

This study investigates the comparative effect of UF profiling versus non-profiled conventional HD on select cardiovascular and patient-reported outcomes. Participants will complete two phases of UF profiling and two phases of conventional HD and will act as their own controls.

ELIGIBILITY:
Inclusion Criteria:

* UF rate >10 mL/h/kg in >30% of treatments in a 30-day screening period (require ≥6 outpatient HD treatments in this period)
* Age 18-85 years
* Ability to converse comfortably in English or Spanish
* Receipt of in-center maintenance HD at Carolina Dialysis clinics in Carrboro or Siler City, North Carolina
* ≥90 days on HD
* Free of bloodstream infection during screening period
* Willingness to undergo all study testing
* Evidence of a signed and dated informed consent document

Exclusion Criteria:

* Systolic BP unable to be measured by arm cuff
* >1 hospitalization during screening period
* Unstable angina per treating nephrologist
* End-stage cirrhosis per treating nephrologist
* New York Heart Association class IV heart failure per treating nephrologist
* Pregnant
* More than 4 times per week HD
* Incarcerated
* Anticipated kidney transplant within 6 months per treating nephrologist
* Non-adherence to HD prescription (>2 unexplained absences during screening period)
* Sodium profiling or UF profiling in standard HD prescription
* Decisionally challenged, unable to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Flythe, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Carolina Dialysis - Carrboro, Carrboro, North Carolina
  - Carolina Dialysis - Siler City, Siler City, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flythe JE, Tugman MJ, Narendra JH, Assimon MM, Li Q, Wang Y, Brunelli SM, Hinderliter AL. Effect of ultrafiltration profiling on outcomes among maintenance hemodialysis patients: a pilot randomized crossover trial. J Nephrol. 2021 Feb;34(1):113-123. doi: 10.1007/s40620-020-00862-6. Epub 2020 Sep 25. PMID 32975783

RESULTS

PARTICIPANT FLOW:
Period: Phase 1 Intervention (3 Weeks)
Arm/Group | UF Profiling Phase First | Conventional HD Phase First
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0
Period: First Washout (1 Week)
Arm/Group | UF Profiling Phase First | Conventional HD Phase First
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0
Period: Phase 2 Intervention (3 Weeks)
Arm/Group | UF Profiling Phase First | Conventional HD Phase First
Started | 18 | 16
Completed | 17 | 16
Not Completed | 1 | 0
Not completed — Kidney Transplant | 1 | 0
Period: Second Washout (1 Week)
Arm/Group | UF Profiling Phase First | Conventional HD Phase First
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0
Period: Phase 3 Intervention (3 Weeks)
Arm/Group | UF Profiling Phase First | Conventional HD Phase First
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0
Period: Third Washout (1 Week)
Arm/Group | UF Profiling Phase First | Conventional HD Phase First
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0
Period: Phase 4 Intervention (3 Weeks)
Arm/Group | UF Profiling Phase First | Conventional HD Phase First
Started | 17 | 16
Completed | 16 | 16
Not Completed | 1 | 0
Not completed — Prolonged Hospitalization | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UF Profiling Phase First | Conventional HD Phase First | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55 (15) | 57 (15) | 56 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 10 | 22
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Intradialytic Hypotension (Intradialytic Hypotension Defined as Nadir Systolic BP <90 mmHg)
Description: Intradialytic blood pressure (BP) was measured with an upper extremity cuff in seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Intradialytic hypotension was defined as the presence of a nadir systolic BP <90 mmHg. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Every study hemodialysis treatment, up to 36 treatments per participant over 15 weeks
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Groups:
- UF Profiling: Linear UF profiling (linearly decreasing UF rate with a UF rate starting at 1.33 times the rate that would be needed at a constant UF rate to achieve the desired post-weight; preprogrammed "profile 2" on a Fresenius 2008K machine). Ultrafiltration profiling performed using Fresenius 2008K dialysis machines in accordance with manufacturer instructions.
- Conventional HD: Conventional HD (routine care) is the participant's standard HD prescription without UF profiling
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 578 | 571
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in intradialytic hypotension between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — The equivalence margin is the standard error of the estimated differences between UF and standard treatment from the repeated measure mixed model; p = 0.5, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.8 to 1.7]

2. Primary Outcome: Pre- to Post-hemodialysis Treatment Change in Troponin T Level in ng/mL at Weeks 3, 7, 11, and 15, Using Mixed Model Analysis
Description: Troponin T blood samples were collected at 4 study visits. Specifically, at the 7th hemodialysis treatment in each respective study phase (i.e., at week 3, 7, 11, and 15 study visits). Pre- to post-hemodialysis troponin T change was calculated as: post-dialysis troponin T - pre-dialysis troponin T (ng/mL). A lower change value reflects less cardiac strain. Based on the pre-specified protocol, the reported values represent change in troponin T between pre- and post-hemodialysis using mixed model (repeated measures logistic regression) analysis that considered all specified time-points (i.e., weeks 3, 7, 11, and 15).
Time Frame: Weeks 3, 7, 11, and 15
Population: All participants who completed at least one phase of each study arm.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
ng/mL | 12.3 [4.4 to 20.2] | 11.3 [3.4 to 19.2]
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in troponin T change between UF profiling and conventional HD. Repeated measure linear regression was performed, giving each subject a random intercept term. The coefficient is the difference in the outcome between UF profiling and conventional HD; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.2, Mixed Models Analysis — Statistically significant p-value is <0.05; Beta coefficient = -2.8, 95% CI 2-sided [-6.9 to 1.4]

3. Primary Outcome: Occurrence of a ≥10% Troponin T Percentage Rise From Pre- to Post-hemodialysis Treatment
Description: Troponin T blood samples were collected before and after each participant's 7th hemodialysis treatment of each study phase (4 times during the study). Troponin T percentage change was calculated as [(Post-HD troponin T - pre-HD troponin T) / pre-HD troponin T] x100. Troponin T percentage rise was defined as a troponin T percentage change ≥10%. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 3, 7, 11, and 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 64 | 63
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in troponin T rise between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.2 to 1.3]

4. Primary Outcome: Change From Baseline in Percent Left Ventricular Global Longitudinal Strain (GLS)
Description: Left ventricular GLS was measured with transthoracic echocardiography at baseline and at 30 minutes before HD treatment end during the 7th treatment in the first phase of each arm. Left ventricular GLS change was calculated as peak intradialytic stress GLS - baseline GLS (%). A lower change value reflects lesser cardiac strain. Median differences were estimated using Wilcoxon (Mann-Whitney) tests.
Time Frame: Weeks 3 and 7
Population: All participants who had baseline GLS measurement and had one GLS measurement in each study arm.
Measure: Median (95% Confidence Interval); unit: GLS change (%)
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 29 | 27
GLS change (%) | 0.9 [-0.1 to 1.8] | 1.3 [0.1 to 2.4]
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in left ventricular GLS change between UF profiling and conventional HD. Wilcoxon (Mann-Whitney) tests were performed assessing the difference of the endpoint between the 2 treatment groups; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.2, Wilcoxon (Mann-Whitney) — Statistically significant p-value is <0.05; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.0 to 0.5]

5. Secondary Outcome: Nadir Systolic Blood Pressure During Hemodialysis in mmHg
Description: Intradialytic BP was measured with an upper extremity cuff in seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Nadir systolic BP was defined as the lowest intradialytic systolic BP measurement during each hemodialysis treatment. Lower values reflect greater cardiac strain. Beta-coefficients were estimated using a mixed model (repeated measures linear regression model).
Time Frame: Every study hemodialysis treatment, up to 36 treatments per participant over 15 weeks
Population: All participants who completed at least one phase of each study arm.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
mmHg | 104.9 [98.4 to 111.4] | 102.1 [95.5 to 108.6]
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in nadir systolic BP between UF profiling and conventional HD. Repeated measure linear regression was performed, giving each subject a random intercept term. The coefficient is the difference in the outcome between UF profiling and conventional HD; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9, Mixed Models Analysis — Statistically significant p-value is <0.05; Beta coefficient = -0.2, 95% CI 2-sided [-2.0 to 1.7]

6. Secondary Outcome: Occurrence of Failed Target Weight Achievement (Failed Target Weight Achievement Defined as a Difference in Prescribed Target Weight and Post-dialysis Weight That is >1 kg or <-1 kg)
Description: The treating nephrologist prescribed the target weight per routine clinical care. Post-dialysis weight was measured after each hemodialysis treatment in the standing position, per dialysis clinic protocol. Failed target weight achievement was defined as a difference in prescribed target weight and post-dialysis weight that was >1 kg or <-1 kg. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Every study hemodialysis treatment, up to 36 treatments per participant over 15 weeks
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 578 | 571
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in failed target weight achievement between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.8, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.7 to 1.3]

7. Secondary Outcome: Occurrence of Patient-reported Clinically Important Cramping During Dialysis (Clinically Important Cramping Defined as Moderate, Severe, or Very Severe Cramping)
Description: Participants' dialysis-related symptoms (e.g. cramping) during the last week were assessed using an investigator-developed 12-question symptom questionnaire administered once weekly throughout the study (6 times per study arm). Each symptom was graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Clinically important cramping was defined as cramping ranked as moderate, severe or very severe. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 1, 2, 3, 5, 6, 7, 9, 10, 11, 13, 14, 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 245 | 242
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in clinically important cramping between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.9, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.4 to 2.1]

8. Secondary Outcome: Occurrence of Patient-reported Clinically Important Nausea or Upset Stomach During Dialysis (Clinically Important Nausea or Upset Stomach Defined as Moderate, Severe, or Very Severe Nausea or Upset Stomach)
Description: Participants' dialysis-related symptoms (e.g. nausea or upset stomach) during the last week were assessed using an investigator-developed 12-question symptom questionnaire administered once weekly throughout the study (6 times per study arm). Each symptom was graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Clinically important nausea/upset stomach was defined as nausea/upset stomach ranked as moderate, severe or very severe. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 1, 2, 3, 5, 6, 7, 9, 10, 11, 13, 14, 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 245 | 242
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in clinically important nausea/upset stomach between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.5, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.2 to 2.2]

9. Secondary Outcome: Occurrence of Patient-reported Clinically Important Vomiting or Throwing up During Dialysis (Clinically Important Vomiting or Throwing up Defined as Moderate, Severe, or Very Severe Vomiting or Throwing up)
Description: Participants' dialysis-related symptoms (e.g. vomiting or throwing up) during the last week were assessed using an investigator-developed 12-question symptom questionnaire administered once weekly throughout the study (6 times per study arm). Each symptom was graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Clinically important vomiting/throwing up was defined as vomiting/throwing up ranked as moderate, severe or very severe. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 1, 2, 3, 5, 6, 7, 9, 10, 11, 13, 14, 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 245 | 242
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in clinically important Vomiting/throwing up score between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0, Mixed Models Analysis; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.1 to 16.0]

10. Secondary Outcome: Occurrence of Patient-reported Clinically Important Dizziness or Lightheadedness During Dialysis (Clinically Important Dizziness or Lightheadedness Defined as Moderate, Severe, or Very Severe Dizziness or Lightheadedness)
Description: Participants' dialysis-related symptoms (e.g. dizziness or lightheadedness) during the last week were assessed using an investigator-developed 12-question symptom questionnaire administered once weekly throughout the study (6 times per study arm). Each symptom was graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Clinically important dizziness/lightheadedness was defined as dizziness/lightheadedness ranked as moderate, severe or very severe. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 1, 2, 3, 5, 6, 7, 9, 10, 11, 13, 14, 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 245 | 242
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in clinically important dizziness/lightheadedness between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.04, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 0.2, 95% CI 2-sided [0.1 to 0.9]

11. Secondary Outcome: Occurrence of Patient-reported Clinically Important Racing Heart or Heart Palpitations During Dialysis (Clinically Important Racing Heart or Heart Palpitations Defined as Moderate, Severe, or Very Severe Racing Heart or Heart Palpitations)
Description: Participants' dialysis-related symptoms (e.g. racing heart or heart palpitations) during the last week were assessed using an investigator-developed 12-question symptom questionnaire administered once weekly throughout the study (6 times per study arm). Each symptom was graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Clinically important racing heart/heart palpitations was defined as racing heart/heart palpitations ranked as moderate, severe or very severe. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 1, 2, 3, 5, 6, 7, 9, 10, 11, 13, 14, 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 245 | 242
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in clinically important racing heart/heart palpitations between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.3, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 3.1, 95% CI 2-sided [0.3 to 32.4]

12. Secondary Outcome: Occurrence of Patient-reported Clinically Important Chest Pain During Dialysis (Clinically Important Chest Pain Defined as Moderate, Severe, or Very Severe Chest Pain)
Description: Participants' dialysis-related symptoms (e.g. chest pain) during the last week were assessed using an investigator-developed 12-question symptom questionnaire administered once weekly throughout the study (6 times per study arm). Each symptom was graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Clinically important chest pain was defined as chest pain ranked as moderate, severe or very severe. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 1, 2, 3, 5, 6, 7, 9, 10, 11, 13, 14, 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 245 | 242
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in clinically important chest pain between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.0, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.2 to 6.0]

13. Secondary Outcome: Occurrence of Patient-reported Clinically Important Shortness of Breath During Dialysis (Clinically Important Shortness of Breath Defined as Moderate, Severe, or Very Severe Shortness of Breath)
Description: Participants' dialysis-related symptoms (e.g. shortness of breath) during the last week were assessed using an investigator-developed 12-question symptom questionnaire administered once weekly throughout the study (6 times per study arm). Each symptom was graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Clinically important shortness of breath was defined as shortness of breath ranked as moderate, severe or very severe. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 1, 2, 3, 5, 6, 7, 9, 10, 11, 13, 14, 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 245 | 242
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in clinically important shortness of breath between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.7, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.3 to 6.5]

14. Secondary Outcome: Occurrence of Patient-reported Clinically Important Thirst or Dry Mouth During Dialysis (Clinically Important Thirst or Dry Mouth Defined as Moderate, Severe, or Very Severe Thirst or Dry Mouth)
Description: Participants' dialysis-related symptoms (e.g. thirst or dry mouth) during the last week were assessed using an investigator-developed 12-question symptom questionnaire administered once weekly throughout the study (6 times per study arm). Each symptom was graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Clinically important thirst/dry mouth was defined as thirst/dry mouth ranked as moderate, severe or very severe. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 1, 2, 3, 5, 6, 7, 9, 10, 11, 13, 14, 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 245 | 242
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in clinically important thirst/dry mouth between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.2, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.3 to 1.2]

15. Secondary Outcome: Occurrence of Patient-reported Clinically Important Headache During Dialysis (Clinically Important Headache Defined as Moderate, Severe, or Very Severe Headache)
Description: Participants' dialysis-related symptoms (e.g. headache) during the last week were assessed using an investigator-developed 12-question symptom questionnaire administered once weekly throughout the study (6 times per study arm). Each symptom was graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Clinically important headache was defined as headache ranked as moderate, severe or very severe. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 1, 2, 3, 5, 6, 7, 9, 10, 11, 13, 14, 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 245 | 242
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in clinically important headache between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.8, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.4 to 2.3]

16. Secondary Outcome: Occurrence of Patient-reported Clinically Important Itching During Dialysis (Clinically Important Itching Defined as Moderate, Severe, or Very Severe Itching)
Description: Participants' dialysis-related symptoms (e.g. itching) during the last week were assessed using an investigator-developed 12-question symptom questionnaire administered once weekly throughout the study (6 times per study arm). Each symptom was graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Clinically important itching was defined as itching ranked as moderate, severe or very severe. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 1, 2, 3, 5, 6, 7, 9, 10, 11, 13, 14, 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 245 | 242
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in clinically important itching between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.02, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 2.8, 95% CI 2-sided [1.2 to 6.6]

17. Secondary Outcome: Occurrence of Patient-reported Clinically Important Restless Legs During Dialysis (Clinically Important Restless Legs Defined as Moderate, Severe, or Very Severe Restless Legs)
Description: Participants' dialysis-related symptoms (e.g. restless legs) during the last week were assessed using an investigator-developed 12-question symptom questionnaire administered once weekly throughout the study (6 times per study arm). Each symptom was graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Clinically important restless legs was defined as restless legs ranked as moderate, severe or very severe. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 1, 2, 3, 5, 6, 7, 9, 10, 11, 13, 14, 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 245 | 242
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in clinically important restless legs/difficulty keeping legs still between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.7, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.5 to 2.6]

18. Secondary Outcome: Occurrence of Patient-reported Clinically Important Tingling or Feeling of Pins and Needles During Dialysis (Clinically Important Tingling or Feeling of Pins and Needles Defined as Moderate, Severe, or Very Severe Tingling or Feeling of Pins and Needles)
Description: Participants' dialysis-related symptoms (e.g. tingling or feeling of pins and needles during the last week were assessed using an investigator-developed 12-question symptom questionnaire administered once weekly throughout the study (6 times per study arm). Each symptom was graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Clinically important tingling/feeling of pins and needles was defined as tingling/feeling of pins and needles ranked as moderate, severe or very severe. Odds ratios were estimated using a mixed model (repeated measures logistic regression model).
Time Frame: Weeks 1, 2, 3, 5, 6, 7, 9, 10, 11, 13, 14, 15
Population: All participants who completed at least one phase of each study arm.
Measure: Number; unit: Number of occurrences
Arm/Group | UF Profiling | Conventional HD
Number analyzed (Participants) | 33 | 33
Number of occurrences | 245 | 242
Statistical Analysis 1: Comparison: UF Profiling vs Conventional HD; Null hypothesis = no difference in clinically important tingling/feeling of pins and needles between UF profiling and conventional HD. Likelihood ratio tests were performed using repeated measure logistic regression with the binary treatment indicator as a fixed effect predictor and assigning each subject a random intercept term. A likelihood ratio test assessed the significance of whether the coefficient corresponding to the binary treatment indicator equals to zero; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.5, Mixed Models Analysis — Statistically significant p-value is <0.05; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.2 to 2.4]

ADVERSE EVENTS:
Time Frame: From the time informed consent is obtained to study participation end, up to 21 weeks.
Arm/Group | UF Profiling | Conventional HD
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 2/34 | 5/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UF Profiling (N=34) | Conventional HD (N=34)
Epistaxis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Missed study treatment due to hospitalization
Clostridium difficile diarrhea (Infections and infestations) | 1 (1) | 0 (0) — Missed study treatment due to hospitalization
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) — Missed study treatment due to hospitalization
Hypervolemia (Cardiac disorders) | 0 (0) | 1 (2) — Missed study treatment due to hospitalization
Arteriovenous vascular access surgery (Surgical and medical procedures) | 0 (0) | 1 (3) — Missed study treatment due to hospitalization
Bone fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (8) — Missed study treatment due to hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT03301740/Prot_SAP_000.pdf